CLINICAL TRIAL: NCT02189460
Title: Cognitive Mechanisms and Cerebral Substrate of Naming Impairment During Aging. Behavior and Neuroimaging Approaches.
Brief Title: Effect of Normal Aging on Language Processing
Acronym: SEMVIE
Status: Terminated | Type: Observational
Why Stopped: Not enough subjects
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-AZ00569-38
Record Dates: First submitted 2014-07-03; First posted 2014-07-14 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Cognition
Keywords: Cognition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy adults: 20 young adults aged between 30 and 50 years old. 20 middle aged adults aged between 50 and 70 years old. 20 older adults of 70 years old and more.

SUMMARY:
The purpose of this study is to understand the effect of age on language abilities. The investigators aim at investigating the cerebral modifications that take place in normal aging, at the functional an anatomical level.

ELIGIBILITY:
Inclusion Criteria:

* Age of 30 years and above
* Right handed
* French native speakers
* Affiliation to French social security (Sécurité Sociale)
* Medical interview
* Consent form signed

Exclusion Criteria:

* Cerebral or respiratory pathologies
* Any MRI contrindication

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 healthy adults will participate to the study. There will be 3 age groups: 30-50, 50-70, > 70 years. Ech group will contain 20 volunteers.
  The volunteers are recruited by means of ads on Laboratory websites and Universities.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-07; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent functional MRI | There will be a unique MRI measurement for each participant. Group analyses presentation after 1 year.
  We use 3 functional tasks using block paradigm: Object naming, Verbal generation and semantic judgment, to elicit BOLD response using fMRI in order to compare functional activation patterns between subjects.
  We also use hypercapnic challenge to elicit BOLD response in order to obtain Cerebral Vascular Reactivity properties of subjects.
Anatomical MRI | There will be a unique MRI measurement for each participant. Group analyses presentation after 1 year.
  We use Voxel Based Morphometry to compare cortical volume (grey matter) between subjects.
  We also use tractography Diffusion Tensor Imaging to compare white matter properties between subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Krainik, Professor, Principal Investigator — Neuroradiology department, Grenoble Hospital, INSERM, Grenoble University.; Monica Baciu, Professor, Study Director — Laboratory of Psychology and NeuroCognition, CNRS, Grenoble University.
Locations (1):
- IRMaGe facility, Grenoble, France